CLINICAL TRIAL: NCT03289390
Title: Treatment of a PDA With Acetaminophen in Preterm Neonates: Exploring Various Indications
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Ronnelle King, MD, Albany Medical College
Other Study IDs: 4846
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acetaminophen to close PDA: Infants with PDA treated with acetaminophen beyond 14 days of life or in whom acetaminophen is used due to contraindication to ibuprofen
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen given at discretion of medical team for PDA treatment. Research team to evaluate pre and post laboratory values and echocardiograms.

SUMMARY:
This study will evaluate the use of acetaminophen in preterm infants when a patent ductus arteriosus (PDA) is of concern. We will perform two simultaneous prospective observational studies over a 3 year period. The first will be of infants with clinically significant PDAs beyond 14 days of life who are medically treated with acetaminophen as a means to avoid surgical ligation, and the second will be of infants who received acetaminophen for a PDA closure during the first 2 weeks of life as a result of ibuprofen, the current standard of care in our NICU, contraindication due to medical status.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 23 0/7 to 29 6/7 weeks gestation, with PDA determined by medical team to need treatment and infant is beyond 14 days of life.

Exclusion Criteria:

* Congenital heart disease Pneumonia Pulmonary hypertension Pulmonary hemorrhage ALT and AST ≥ 2X the upper limit of normal (=AST> 150 U/L, ALT>90 U/L) Sepsis/meningitis Abnormal chromosomes Hydrops Major congenital malformations

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants born between 23 0/7 weeks to 29 6/7 weeks gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of PDA closure | 3 days
  PDA will be evaluated by echocardiography to determined whether it has closed after treatment is complete.
Change in PDA size | 3 days
  Size of PDA will be measured by echocardiography to determine if the size has changed after treatment is complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Mashad AE, El-Mahdy H, El Amrousy D, Elgendy M. Comparative study of the efficacy and safety of paracetamol, ibuprofen, and indomethacin in closure of patent ductus arteriosus in preterm neonates. Eur J Pediatr. 2017 Feb;176(2):233-240. doi: 10.1007/s00431-016-2830-7. Epub 2016 Dec 21. PMID 28004188
- [Background] EL-Khuffash A, James AT, Cleary A, Semberova J, Franklin O, Miletin J. Late medical therapy of patent ductus arteriosus using intravenous paracetamol. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F253-6. doi: 10.1136/archdischild-2014-307930. Epub 2015 Feb 4. PMID 25653299